CLINICAL TRIAL: NCT07070245
Title: Comparing Instrument Assisted Soft Tissue Mobilization With Positional Release Technique for Plantar Fasciitis Pain and Range of Motion
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Doaa Said Mohamed Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Doaa Said Mohamed Ibrahim, Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No:P.T.REC/012/005492
Record Dates: First submitted 2025-07-05; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Plantar Fasciitis; Heel Pain; Plantar Fascia Inflammation
Keywords: Instrument assisted soft tissue mobilization; Chronic plantar fasciitis; Positional release technique
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positional release technique (Experimental): Positional release technique in addition to exercises in form of stretching exercises for plantar fascia, gastrocnemius, soleus muscles, and short foot exercise (study group) The treatment protocol will be two sessions. given per week for 4 weeks.
  Interventions: Procedure: Positional release
- Traditional exercises (control group) (Experimental): Traditional exercises (control group), traditional exercises in form of stretching exercises for plantar fascia, gastrocnemius, soleus muscles, and short foot exercise The treatment protocol will be two sessions.
  given per week for 4 weeks.
  Interventions: Procedure: Exercises
- Instrument assisted soft tissue mobilization (Experimental): Instrument-assisted soft tissue mobilization in addition to exercises (study group) in form of stretching exercises for plantar fascia, gastrocnemius, soleus muscles, and short foot exercise
  Interventions: Procedure: Instrument assisted soft tissue mobilization

INTERVENTIONS:
Procedure: Instrument assisted soft tissue mobilization — The treatment protocol will be two sessions. given per week for 4 weeks.
  Arms: Instrument assisted soft tissue mobilization
Procedure: Positional release — The treatment protocol will be two sessions. given per week for 4 weeks.
  Arms: Positional release technique
Procedure: Exercises — The treatment protocol will be two sessions. given per week for 4 weeks.
  Arms: Traditional exercises (control group)

SUMMARY:
Chronic plantar fasciitis (CPF) is the most common cause of chronic heel pain in adults, affecting both young active patients and older, more sedentary individuals. It results from chronic overload of the plantar fascia. This overload may be due to overuse, as seen in runners and military personnel, or due to excessive loading in individuals with obesity (body mass index >30), sedentary lifestyles, or occupations that require prolonged standing.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed cases of plantar fasciitis not less than 3 months.
2. Heel pain felt maximally over plantar aspect of heel.
3. Pain in the heel on the first step in the morning.
4. Their age ranging from 30 to 50 years

Exclusion Criteria:

1. Subjects can't tolerate close physical contact (Kotwalkar et al., 2019).
2. Athletes.
3. Subjects with skin infections (Kotwalkar et al., 2019).
4. Subjects with recent fracture with incomplete bony union (Rowlett et al., 2018).
5. Subjects with acute inflammatory or infectious process (Rowlett et al., 2018).
6. Subjects with hematoma (Rowlett et al., 2018).
7. Subjects with osteoporosis (Looney et al., 2011).
8. Subjects with foot deformity (Kotwalkar et al., 2019).
9. Subjects that take medications that may increase blood clotting (Kotwalkar et al., 2019).
10. Surgery to the ankle or foot (Looney et al., 2011).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-22 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity level assessed by Numeric Pain Rating Scale (NPRS) | Baseline and after 8 sessions (approximately 4 weeks)
  Pain intensity level assessed by Numeric Pain Rating Scale. A scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
Range of motion | Baseline and after 8 sessions (approximately 4 weeks)
  A digital goniometer is used for the assessment of ankle dorsiflexion, plantar flexion range of motion, and knee flexion range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Port Said, Port Said Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and limitations in data-sharing agreements.

REFERENCES:
- [Background] Neufeld SK, Cerrato R. Plantar fasciitis: evaluation and treatment. J Am Acad Orthop Surg. 2008 Jun;16(6):338-46. doi: 10.5435/00124635-200806000-00006. PMID 18524985